CLINICAL TRIAL: NCT04541940
Title: TeleRehabilitation Following ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-01260
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Active Comparator)
  Interventions: Other: Telerehabilitation Therapy
- In-Person Rehabilitation (Active Comparator)
  Interventions: Other: In-person Rehabilitation Therapy

INTERVENTIONS:
Other: Telerehabilitation Therapy — Rehabilitation services will be dispensed at patients' home utilizing video telecommunication services with real-time synchronous exchange of information - Quadriceps isometrics exercises, straight leg raises, and range of motion exercises.
  Arms: Telerehabilitation
Other: In-person Rehabilitation Therapy — Quadriceps isometrics exercises, straight leg raises, and range of motion exercises.
  Arms: In-Person Rehabilitation

SUMMARY:
Telerehabilitation is a form of tele-treatment in which rehabilitation services are dispensed at patients' home utilizing video telecommunication services with real-time synchronous exchange of information. The advantages of telerehabilitation include reducing unnecessary travel to the hospital and person to person contact while maintaining social distancing. While some of the patients are truly staying at remote areas, others are unable to manage travel in the lockdown period. Telemedicine offers the opportunity to deliver rehabilitative services in the patients' home, closing geographic, physical, and motivational gaps. Punctuality on either side is also assured since the travel times are saved on both the ends.

The purpose of the proposed study is to evaluate telerehabilitation vs. in-person rehabilitation following ACL reconstruction. Objectives include assess return to sport and patient reported functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for ACL reconstruction
* Age 18-40
* Ability to comply with a standardized postoperative protocol
* Willing and able to provide consent

Exclusion Criteria:

* Pregnant patient
* Age >40 years, or < 18
* Previous knee surgery
* Unable to speak English or perform informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
RTS (Return to Sport) | up to 1 year post-op
  The day when the participant is able to fully participate in their sport, but not at their desired performance level.

SECONDARY OUTCOMES:
ACL-RSI Questionnaire Score | up to 1 year post-op
  ACL-RSI (anterior cruciate ligament - return to sport) consists of 12 questions. Each question is scored 0-100 with a total range of 0-1200. The higher the score, the more positive psychological outlook a participant has.
Visual Analogue Scale (VAS) Score | up to 1 year post-op
  VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The total score ranges from 0-10. The higher the score, the worse the pain.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | up to 1 year post-op
  KOOS is a knee-specific instrument, developed to assess the participants' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales. Each subscale is calculated independently. The calculated mean score of the individual items of each subscale will be divided by 4. The total score range is 0-100. The lower the score, the more extreme the problems.
International Knee Documentation Committee (IKDC) Score | up to 1 year post-op
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Campbell, MD, Principal Investigator — kirk.campbell@nyulangone.org
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to kirk.campbell@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.